CLINICAL TRIAL: NCT04327128
Title: Evaluation of a Digital Support and Communication Platform for Heart Failure:
Brief Title: Selfcare MAnagement InteRvenTion in Heart Failure II (SMART HF II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Sofia Gerward, Principal Investigator, Lund University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SMART HF II, Dnr 20 19-00378
Record Dates: First submitted 2020-03-15; First posted 2020-03-30 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Standard heart failure care and a digital heart failure support system
  Interventions: Device: LifePod
- Control group (Other): Standard heart failure care
  Interventions: Device: LifePod

INTERVENTIONS:
Device: LifePod — The intervention group is testing LifePod on a digital communication platform between patient and healthcare provider

SUMMARY:
The purpose of the study is to evaluate if the digital support and communication platform for heart failure can provide patients with heart failure increased knowledge, compliance and quality of life and thus affect re-admissions and visit structure.

To evaluate whether a digital support and communication platform for heart failure patients after 6 months can provide:

1. Improved self-care
2. Improved quality of life and reduced number of patient-assessed symptoms
3. Reduction in the number of cardiovascular events, hospital nights, the number of hospitalizations or the number of deaths and out-patient visits

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed heart failure I.50 (newly discovered or existing) in NYHA Class I-IV in principle with ESC guidelines 2016.

  * Have completed the "consent form" or consent form, see §4.2 Exclusion criteria: * Patient who refuses to participate in the trial.
  * It is assessed that they can handle the intervention themselves or with the help of personal or relatives.

Exclusion Criteria:

* Patient who declines to participate in the trial.

  * Impaired cognitive ability that is judged to affect the ability to conduct the study in the intended manner.
  * Life expectancy <8 months
  * In other ways, by the treating physician, it is deemed inappropriate to participate in the study, e.g. due to participation in another study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Self-care behaviour | 6 month
  Improvement in self-care behaviour measured by the questionnaire European Heart Failure Self-care behaviour scale (EHFScB-9) A higher EHFScB-9 score indicates a worse self-care behaviour. The minimum score is 9 points and the maximum score is 45.
Cardiovascular events and deaths | 12 month
  Number of participants with cardiovascular events and deaths during intervention and up to 12 months after inclusion
Hospitalization and hospital days | 12 months
  Number of participants with new hospitalization and number of hospital days during intervention and up 12 months after inclusion
Health care visits | 12 months
  Type and number of health care visits during intervention and up to 12 months after inclusion
Patient-reported symptoms | 6 months
  Improved patient-reported symptoms as measured by questionnaire EuroQol three-dimensional questionnaire (EQ-5D-3L ) where high score represent worse symptoms. The minimum score is 7 points and the maximum score is 23 points.
Quality of life | 6 months
  Improved quality of life as measured on visual analogue scale 0-100 where high figure represent best quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Gerward, MD, PhD, Principal Investigator — Lund University
Locations (1):
- Lund University, Lund, Skåne County, Sweden